CLINICAL TRIAL: NCT05402228
Title: Investigation of the Aural Symptoms and Dizziness in Patients With Temporomandibular Joint Disorders
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Medical Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2022.03.55
Record Dates: First submitted 2022-05-28; First posted 2022-06-02 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Temporomandibular Joint Disorders; Dizziness; Tinnitus
Keywords: temporomandibular joint; dizziness; aural sypmtoms; tinnitus
MeSH Terms: conditions — Temporomandibular Joint Disorders; Dizziness; Tinnitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: temporomandbular joint disorders — no intervention

SUMMARY:
120 male and female patients aged between 18-65 years who apply to the outpatient clinic and diagnosed with TMD will be included in the study. Patients will be divided into 3 groups as Muscle Disorders (Group 1), Temporomandibular Joint Disorders (Group 2) and degenerative joint diseas (osteoarthrosis) (Group 3) according to DC/TMD axis I diagnostic criteria.

maximum mouth opening, TMJ sound, pain levels, tinnitus, and dizziness are evaluated.

DETAILED DESCRIPTION:
120 male and female patients aged between 18-65 years who apply to the outpatient clinic and diagnosed with TMD will be included in the study. Patients will be divided into 3 groups as Muscle Disorders (Group 1), Temporomandibular Joint Disorders (Group 2) and degenerative joint diseas (osteoarthrosis) (Group 3) according to DC/TMD axis I diagnostic criteria.

Demographic data of all patients participating in the study will be obtained. Then, physical examination will reveal maximum mouth opening, right and left lateral movement, deflexion, deviation. Accompanying tinnitus, ear fullness and dizziness will be questioned.

All measurements, including maximum mouth opening, and physical examination will be performed with patients sitting upright in an anatomical position in a chair. All measurements will be performed by the same physical therapist with 7 years of experience in TMD.

In the measurement of maximum mouth opening, patients will be asked to open their mouths as wide as possible. The distance between the anterior incisors is measured with the help of a ruler suitable for millimeter measurement. Maximum mouth opening distance is a physical examination method frequently used to determine the motion and function of the jaw joint. Functional mouth opening is accepted as 35-40 mm (12).

For the evaluation of TMJ sound, the TMJ is palpated with the thumb and middle fingers and the sound heard when opening and closing the mesh is noted.

Pain levels are measured using a 10-point visual analog scale (VAS). The presence of bruxism is determined on physical examination based on the presence of abnormal tooth wear, tooth marks in the buccal region, tooth marks on the tongue, and hypertrophy of the masseter muscle.

The sense of fullness in the ear, tinnitus, and dizzyness, which the patients reported themselves, is questioned. The relationship between having TMD, clinical characteristics and dizziness will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* being 18-65 years of age
* diagnosed with TMD

Exclusion Criteria:

* Lack of cognitive ability to understand test instructions, illliteracy, aphasia, presence of a known psychiatric illness
* Patients under the age of 18 and over the age of 65
* Having another systemic disease that will cause TMD (cancer, rheumatological diseases)
* Presence of disease that will increase a anotherural symptoms or cause d d (presence of disease of vertigo, history of vertigo)
* Presence of a history of cervical pain, cervical spondylosis, cervical disc herniation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants aged 18-65 years with TMD
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
maximum mouth opening | 1 day
  maximum mouth opening
right and left lateral movement, deflexion, and deviation | 1 day
  right and left lateral movement, deflexion, and deviation
TMJ sound | 1 day
  the TMJis palpated with the thumb and middle fingers and the sound heard when opening and closing the mesh was noted.
visual analog scale | 1 day
  It is use for evaluate the pain intensity.

SECONDARY OUTCOMES:
bruxism | 1 day
  it is determined on physical examination based on the presence of abnormal tooth wear, tooth marks in the buccal region, tooth marks on the tongue, and hypertrophy of the masseter muscle.
the presence of bruxism, tinnitus and dizzeness | 1 day
  the presence of bruxism, tinnitus and dizzeness

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)